CLINICAL TRIAL: NCT05345847
Title: A Study to Evaluate the Efficacy and Safety of Steroid Sparing Strategy in Immune Related Hepatitis
Brief Title: Steroid Sparing in Immune Related Hepatitis (irH)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMPACT 7.0
Record Dates: First submitted 2022-03-23; First posted 2022-04-26 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Hepatitis Immune
Keywords: immune related hepatitis; steroid sparing
MeSH Terms: interventions — Watchful Waiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1- Active Surveillance (Experimental): Active surveillance with rescue corticosteroids
  Interventions: Other: Active Surveillance
- 2- Early initiation of steroid (Standard) (Active Comparator): Early intervention with high-dose steroids
  Interventions: Other: Early initiation

INTERVENTIONS:
Other: Active Surveillance — Close monitoring of liver enzymes with steroid rescue strategy (watch and wait approach)
  Arms: 1- Active Surveillance
Other: Early initiation — Immediate start of high-dose steroids
  Arms: 2- Early initiation of steroid (Standard)

SUMMARY:
A multi-centre, randomized, non-inferiority trial in patients with irH, randomized to receive either close surveillance with corticosteroid rescue therapy or early high dose corticosteroids.

DETAILED DESCRIPTION:
Immune checkpoint inhibitors (ICIs) are a class of immunotherapy drugs that helps signal to the immune system to seek out and destroy cancer. However despite showing clinical benefit over traditional chemotherapy, ICIs can lead to certain toxicities called immune-related adverse events (irAEs).

One of these irAEs is immunotherapy related hepatitis (irH) and is an important and less common toxicity of ICI therapy that could develop into a rare but serious complication of sudden liver failure. The management of irH includes high-dose steroids and use of steroids is not without significant side effects, especially when used for longer term.

Given the potential consequences of high dose long-term corticosteroids along with the implications of permanently discontinuing therapy, it is necessary to better understand the pathophysiology associated with irH and clarify the role of steroids in managing this patient population. It is especially important to determine which patients require intervention with steroids and other immunosuppression versus those that could simply be monitored for spontaneous resolution.

The results of this trial will identify predictors of irH resolution and inform judicious use of corticosteroids and immunosuppressive therapy for this at-risk population.

This study has been designed as a randomized, phase II non-inferiority study to investigate the efficacy of an active surveillance with steroid rescue strategy compared to early initiation of corticosteroids in the setting of irH secondary to ICIs. The study treatment period is 12 weeks with twice weekly liver enzyme function assessments. Once irH has improved to by one CTCAE grade (i.e. grade 3 to 2, or grade 2 to 1), this can be decreased to weekly assessment. For patients who continue to have asymptomatic liver enzyme elevation of grade 2 or higher, maintaining a surveillance strategy beyond this point is not appropriate, as investigators may wish to adjust therapy, especially if this is resulting in delay in resuming ICI. In this setting, weekly liver enzyme assessment will continue. The frequency of liver enzyme monitoring can be increased at the discretion of the investigator or hepatologist.

Following the initial 12-week period, further surveillance with an observation period consisting of every 3 weekly assessments will be completed for a total of 40 weeks (total study duration of 52 weeks). Participants will continue follow up for a total of one year to allow the capture longer term data as well as other endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be 18 years of age, or older on the day of signing informed consent.
2. Patients must be capable of providing consent to enrolment and treatment.
3. Patients with a performance status of ECOG 0-2 will be eligible for enrolment.
4. Patients with histologically confirmed cancer receiving anti-PD1 or anti-PDL1 monoclonal antibody ICI therapy, either alone or in combination with anti-CTLA-4 monoclonal antibody ICI therapy who develop CTCAEv5.0 grade 2 or grade 3 hepatitis that has developed on, or after, ICI therapy and is felt to be treatment related (irH). Patients must be enrolled on trial within 10 days of diagnosis of grade 2 or grade 3 hepatotoxicity.
5. Absence of any condition hampering compliance with the study protocol and follow- up schedule; those conditions should be discussed with the patient before registration in the trial.
6. Assessment by the Roussel Uclaf Causality Assessment Method (RUCAM) ≥6 showing probable relationship between ICI and liver injury (appendix)

Exclusion Criteria:

1. History underlying liver disease, including, but not limited to: hepatitis B, C, autoimmune hepatitis, primary biliary sclerosis, hemochromatosis, primary sclerosis cholangitis, portal vein thrombosis, Budd Chiari syndrome, alcohol induced hepatitis, suspected drug-induced liver injury from other cause (e.g. acetaminophen, antibiotics, statins, methyldopa, non-prescription herbs, see NIH LiverTox website https://livertox.nih.gov for comprehensive list).
2. If undertaken, liver biopsy supporting a cause of liver dysfunction other than irH
3. Patients with an indication for systemic immunosuppressive medications or corticosteroids. Patients with CTCAEv5.0 grade ≥2 irAE's other than irH (ie. colitis, pneumonitis, rash, etc.) are not eligible for trial, with the exception of endocrinopathies that are being treated with hormone replacement alone and not systemic immunosuppressive medications or corticosteroids.
4. Abnormal International Normalization Ratio (INR) at baseline (≥1.5) and bilirubin ≥60, ALT of ≥10X.
5. Previous use of targeted therapies for treatment of malignancy (e.g. BRAF, MEK, EGFR, and VEGF inhibitors) or current treatment with chemotherapy
6. Present use of warfarin.
7. Diagnosis of immunodeficiency.
8. Current use of immunosuppressive medication, EXCEPT for the following: a. intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection); b. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication).
9. Known prior severe hypersensitivity to investigational product or any component in its formulations, including known severe hypersensitivity reactions to monoclonal antibodies (CTCAEv5.0 Grade ≥ 3).
10. Other severe acute or chronic medical conditions including inflammatory bowel disease, immune pneumonitis, pulmonary fibrosis or psychiatric conditions including recent (within the past year) or active suicidal ideation or behavior; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-12-08 (Actual); Primary Completion 2028-02-08 (Estimated); Study Completion 2029-02-08 (Estimated)

PRIMARY OUTCOMES:
Resolution of biochemical abnormalities in grade 2 and grade 3 irH at 12 weeks. | 12 weeks
  The primary objective of this clinical trial is to determine if active surveillance with steroid salvage is a non-inferior strategy in grade 2 and grade 3 irH in patients without evidence of liver dysfunction. Resolution will be defined as improved in irH to grade ≤1. This was chosen as a clinically significant endpoint as it is often used by oncologists to determine if patients may resume ICI therapy. Assessment and grading will be completed by the investigator according to CTCAEv5.0

SECONDARY OUTCOMES:
Safety of Steroid Sparing Strategy | 1 year
  To evaluate the safety of surveillance strategy based on rates of hospitalization, ICU admission, development of clinically significant liver failure (e.g. decompensated hepatic failure) and death.
Total steroid usage | 1 year
  Total steroid usage (defined as the total amount of prednisone or prednisone equivalent in mg required over the study period).
Development of immune related adverse events (irAE's) other than irH. | 1 year
  Defined as the emergence of adverse events that were not present at study baseline that are deemed by the investigator to be related to prior use of immune checkpoint inhibitors. Causality will be investigator assessed and graded according to CTCAEv5.0.
Re-initiation of immune checkpoint inhibitor therapy. | 1 year
  The proportion of patients in each study arm that are re-treated with an immune checkpoint inhibitor.
The time elapsed between randomization and tumor progression (radiographically or clinically) or death from any cause | 1 year
  Progression free survival

CONTACTS AND LOCATIONS:
Overall Officials: Omar Khan, MD, Principal Investigator — AHS Cancer Control Alberta
Locations (1):
- Arthur J.E. Child Comprehensive Cancer Centre, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No